CLINICAL TRIAL: NCT05310851
Title: The Effect Of Oral Motor Stimulation And Nonnutritive Sucking To The Time Of Transition To Oral Nutrition In Preterm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Merve Çakırlı, Principal Investigator, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EskisehirOU-cakirli-1
Record Dates: First submitted 2022-03-17; First posted 2022-04-05 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Preterm; Nutrition Disorder, Infant; Feeding; Difficult, Newborn
Keywords: preterm; oral motor stimulation; non-nutritive sucking; oral nutrition
MeSH Terms: conditions — Premature Birth; Infant Nutrition Disorders

STUDY DESIGN:
Intervention Model Description: There are three groups in our study. One group will be given a pacifier and the other group will be given a 5-minute oral stimulation program. The other group is the control group.
  39 babies will be included, with 13 babies in each group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PIOMI group (Experimental): Infants in the PIOMI group will receive a 5-minute PIOMI 30 minutes before feeding time. PIOMI will be applied once daily for 14 days.
  Interventions: Other: PIOMI and non-nutritive sucking
- Non-nutritive sucking group (Experimental): Infants in the non-nutritive sucking group will receive pacifier 3 minutes before 1 hour any feeding time and, 2 minutes before 10 minutes. Non-nutritive sucking will be applied once daily for 14 days.
  Interventions: Other: PIOMI and non-nutritive sucking
- control group (No Intervention): only feeding follow-up will be done in the infants in the control group.

INTERVENTIONS:
Other: PIOMI and non-nutritive sucking — PIOMI group; The first three minutes of the five minutes include massages aimed at strengthening the cheeks, lips, gums and tongue; the last two minutes consist of non-feeding suction application.
  Infants in the Non-nutritive sucking group will receive pacifier 3 minutes before 1 hour any feeding time and, 2 minutes before 10 minutes.
  Arms: Non-nutritive sucking group; PIOMI group

SUMMARY:
Oral feeding difficulty is one of the problems that preterm infants frequently experience due to poorly developed oral musculature. Sucking and swallowing are present in early fetal life, but sucking-swallowing and swallowing-respiratory coordination are respectively occurs after the 32 and 33-34 gestational week (GA). For this reason, although there are sucking movements in preterm babies with gestational weeks of 31 and below, oral feeding is difficult because adequate coordination cannot be achieved during sucking-swallowing and breathing. Until these structures develop, preterm babies are fed by gavage (nasogastric/orogastric route) in intensive care units. Gavage feeding causes many negativities such as preventing the advantages of oral nutrition and creating an entry route for infectious agents, and the discharge is also delayed. Thus, infants are exposed to adverse intensive care conditions for a longer period of time. For this reason, it is important to ensure the transition to full oral nutrition as soon as possible.

There are various methods that facilitate the transition of infants to oral feeding. Pacifier and oral stimulation applications are some of them. Oral stimulation was first applied by Fucile et al (2002). It is a method consisting of a total of 15 minutes, in which therapeutic touches are made for 12 minutes before feeding, and in the last few minutes, non-nutritive sucking is applied. Later, Lessen thought that this intervention was longer than the fragile preterm babies with a small oral cavity and shortened the duration of the intervention and reformatted it. This intervention, called "Premature Infant Oral Motor Intervention (PIOMI)" (Preterm Infant Oral Motor Intervention), is a 5-minute application consisting of 3 minutes of massage and 2 minutes of non-nutritive sucking. In the literature review, a study comparing oral motor stimulation and pacifier method was reached. However, in this study, unlike our study, a pacifier was applied to one of the groups, a 12-minute stimulation to the second, and a 12-minute stimulation and pacifier to the third. In our study, there are 3 groups. one of the groups a pacifier will be applied to one group and a 5-minute oral stimulation program will be applied to the other group. The third group is the control group.

The aim of the study is to evaluate the effect of pacifier and oral stimulation applied to preterm infants on the transition time to oral feeding.

DETAILED DESCRIPTION:
The infant hospitalized in the intensive care unit will be evaluated primarily in terms of inclusion criteria in the sample group. The baby meeting the criteria will be evaluated by the neonatologist physician and, if appropriate, interviewed with the parents. Parents will be informed about the study and their written consent will be obtained. The group that the baby will be included in will be determined by the randomization method.

"Preterm Baby Information Form" created by the researcher will fill to all infants in the before the intervention. Then, body weight, height and head circumference will be measured and recorded in order to fill in the 1st day anthropometric measurements information in the Preterm baby follow-up form. Then, "Early Nutrition Skills Assessment Tool (EFS-Turkish)" will be applied to evaluate pre-intervention nutrition skills. Then, intervention will be started. Infants in the PIOMI group will receive a 5-minute PIOMI 30 minutes before feeding time. Infants in the non-nutritive sucking group will receive pacifier 3 minutes before 1 hour any feeding time and, 2 minutes before 10 minutes. PIOMI and non-nutritive sucking will be applied once daily for 14 days. only feeding follow-up will be done in the infants in the control group.

"Early Feeding Skills Assessment Tool (EFS-Turkish)" will be re-administered to all babies at the end of the fourteenth day. Nutritional follow-up will be done until the babies are discharged.

In nutritional follow-up will be evaluated time to transition to full oral feeding and how many cc it takes per minute.

ELIGIBILITY:
Inclusion Criteria:

* gestational age of 29-34 weeks
* Vital signs in balance for at least 24 hours,
* 1st and 5th minute APGAR score of 4 and above,
* postnatal 2-5 days
* Babies with written and verbal consent from their parents

Exclusion Criteria:

* Congenital anomaly
* Necrotizing enterocolitis
* Intraventricular Bleeding
* Babies receiving respiratory support other than high-flow nasal cannula
* Babies who developed any complications during the follow-up period after being included in the study group and whose balance status deteriorated

Ages: 2 Days to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 39 (Actual)
Dates: Start 2021-01-10 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-10 (Actual)

PRIMARY OUTCOMES:
Early Nutrition Skills Assessment Tool (The Early Feeding Skills (EFS) Assessment-Turkish) | first day
  It will be used to assess infants' oral feeding skills and readiness during the transition to oral feeding. Infants will be evaluated on the 1st and 14th days using this scale.A low score indicates that she has no nutritional skills, while a high score indicates that she has nutritional skills.
Early Nutrition Skills Assessment Tool (The Early Feeding Skills (EFS) Assessment-Turkish) | 14th day
  It will be used to assess infants' oral feeding skills and readiness during the transition to oral feeding. Infants will be evaluated on the 1st and 14th days using this scale.A low score indicates that she has no nutritional skills, while a high score indicates that she has nutritional skills.
Nutritional follow-up | average of 1 month
  Nutritional follow-up will be carried out from the day of starting the study until discharge.
  Feeding at 12am and 12pm will be taken into account in the nutrition follow-up. At these feeding times;
  - How many cc it oral takes per minute will be recorded.
Nutritional follow-up | average of 1 month
  Feeding babies with only a bottle or breast 8 times in 48 hours indicates that they are on full oral feeding. Dates when infants transition to full oral feeding will be recorded.

SECONDARY OUTCOMES:
rate of body weight gain | first day
  birth weight and weight on the day of started study will be note.
rate of body weight gain | 7th day
  Weight on the 7th day will be note.
rate of body weight gain | 14th day
  Weight on the 14th day will be note.
rate of body weight gain | one day
  weight on the day of discharge will be note.
discharge time | average of 1 month
  The date of infants admission to the intensive care unit and the date of her discharge will be noted.

CONTACTS AND LOCATIONS:
Overall Officials: Merve Cakirli, Principal Investigator — Eskisehir Osmangazi University
Locations (1):
- Eskisehir Osmangazi University, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No